CLINICAL TRIAL: NCT00389311
Title: A Pilot Protocol to Determine the Effects of Chemical and Mechanical Stress on Rectal Permeability as a Surrogate for Toxicity Evaluation of Rectally Applied Microbicides
Brief Title: A Pilot Study for Toxicity Evaluation of HIV Rectal Microbicides
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Craig W. Hendrix, Professor, Department of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CDC 200-2001-08015-02
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: Microbicide; Safety; HIV prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Plasmalyte A; Nonoxynol

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Nonoxynol-9 (Active Comparator): Gynol-II, 2% N-9, 5 mL
  Interventions: Drug: Nonoxynol-9
- Normosol-R (Other): Normosol-R, 5 mL, single administration, negative control
  Interventions: Drug: Normosol-R
- Normosol with simulation, endoscopy and biopsy (Experimental): Normosol-R, 5 mL following simulation, endoscopy and biopsy
  Interventions: Drug: Normosol-R; Procedure: Gastrointestinal instrumentation

INTERVENTIONS:
Drug: Normosol-R
  Arms: Normosol with simulation, endoscopy and biopsy; Normosol-R
Drug: Nonoxynol-9
  Arms: Nonoxynol-9
Procedure: Gastrointestinal instrumentation
  Arms: Normosol with simulation, endoscopy and biopsy

SUMMARY:
The purpose of this study is to determine if detectable changes in permeability of the lining of the colon are caused by either application of HIV microbicide gels or medical procedures, such as flexible sigmoidoscopy.

DETAILED DESCRIPTION:
It is not currently known if procedures used to observe the lining of the distal colon, such as endoscopy with or without pinch biopsy, may cause mucosal trauma and thus alter colonic permeability. Additionally, the application of topical HIV microbicides (to prevent HIV transmission) and shearing forces associated with rectal intercourse might also adversely affect the epithelial layer, and thus alter colonic permeability. In order to appropriately interpret testing of the effects of topical HIV microbicides on the mucosal lining of the distal colon, it is essential to understand whether these procedures themselves, adversely affect the epithelial layer. If changes in permeability can be detected, this method may be developed to help determine microbicide distribution/toxicity in early phase studies, thus improving the selection of candidate microbicides for study in larger scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 21 years of age
* Prior history of receptive anal intercourse (RAI)
* Subjects must have a history of using commercially-available personal lubricants for RAI.
* Ability to provide signed informed consent.
* Willingness to abstain from lubricant use and anal receptive intercourse for 48 hours prior to and 48 hours after Phases A and B.
* Willingness to use a single dose of rectally-applied N-9.

Exclusion Criteria:

* Mental handicap or impaired cognitive performance status as judged by the investigator.
* Coagulation abnormality which would put the subject at risk for bleeding as judged by the Principal Investigator.
* History of anorectal surgery within the last month or the presence of any anorectal disease or condition that in the judgment of the investigator could affect permeability of the rectal mucosa.
* Presence of any painful anorectal conditions or anorectal lesions that would be tender to manipulation.
* History of occupational radiation exposure.
* History of acute or chronic diarrhea defined as three or more loose stools per day.
* History of any allergic response to rectal lubricants.
* History of sleep apnea, or airway problems with previous sedation procedures.
* History of significant adverse reaction to sedation medications.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Intra-subject comparison of urine and plasma concentrations of 99mTc-DTPA | 0-2 hours, 2-4 hours, 4-8 hours, 8-12 hours and 12-24 hours after introduction of the treatment assignment

CONTACTS AND LOCATIONS:
Overall Officials: Edward Fuchs, PA-C, MBA, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Result] Fuchs EJ, Grohskopf LA, Lee LA, Bakshi RP, Hendrix CW. Quantitative assessment of altered rectal mucosal permeability due to rectally applied nonoxynol-9, biopsy, and simulated intercourse. J Infect Dis. 2013 May 1;207(9):1389-96. doi: 10.1093/infdis/jit030. Epub 2013 Jan 16. PMID 23325915